CLINICAL TRIAL: NCT01732666
Title: Effect of Nefopam on Remifentanil Induced Postoperative Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2011-0883
Record Dates: First submitted 2012-11-18; First posted 2012-11-26 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Patients Undergoing Laparoscopic Gastrectomy
Keywords: Opioid-induced hyperalgesia (OIH)
MeSH Terms: interventions — Nefopam; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group L (Placebo Comparator): receives 100 ml of 0.9% saline immediately after anesthesia induction and 0.05µg/kg/min of remifentanil during anesthesia.
  Interventions: Drug: low dose remifentanil
- group H (Placebo Comparator): 100 ml of 0.9% saline immediately after anesthesia induction and 0.3 µg/kg/min of remifentanil during anesthesia.
  Interventions: Drug: high dose remifentanil
- group N (Experimental): 20mg of nefopam mixed in 100 ml of 0.9% saline immediately after anesthesia induction and 0.3 µg/kg/min of remifentanil during anesthesia.
  Interventions: Drug: Nefopam

INTERVENTIONS:
Drug: Nefopam — 20 mg of Nefopam mixed in 100 ml of 0.9% saline IV immediately after induction of anesthesia.
  Arms: group N
Drug: low dose remifentanil — 100 ml of 0.9% saline immediately after anesthesia induction and 0.05µg/kg/min of remifentanil during anesthesia.
  Arms: group L
Drug: high dose remifentanil — 100 ml of 0.9% saline immediately after anesthesia induction and 0.3 µg/kg/min of remifentanil during anesthesia.
  Arms: group H

SUMMARY:
Opioids has been reported to cause hyperalgesia. Opioid induced hyperalgesia (OIH) is defined as paradoxically lowering the threshold of pain after the exposure of opioid. Remifentanil is a short acting opioid that is commonly used during anesthesia and surgery. However, OIH was reported to occur after surgery when large amount of remifentanil was administered. On the other hand, nefopam is a centrally acting, non-opioid analgesic. Nefopam has been reported to have analgesic and anti-hyperalgesic effect.

The investigators hypothesized that nefopam administration could prevent OIH or reduce the severity of OIH. Therefore, the objective of the study is to find out the effect of nefopam on remifentanil induced hyperalgesia in patients undergoing laparoscopic abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing laparoscopic gastrectomy
2. American Society of Anesthesiologists physical status I or II
3. aged from 20 to 65 years

Exclusion Criteria:

1. Past history of chronic pain
2. Drug or alcohol abuse
3. Psychotic disorder
4. Taking analgesics, anti-epileptics, and anti-depressants.
5. Taking opioids within 24 hrs
6. Renal disease
7. Neuromuscular disease.
8. Moderate to severe cardiovascular disease
9. Pregnant or breast-feeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Hyperalgesic extent around surgical incision | Postoperative 24 hr and 48 hr
  The distance from the surgical incision to a point where patient does not feel pain when he gets stimuli with von Frey filament No.16 (122g/mm2).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea